CLINICAL TRIAL: NCT04816071
Title: Essential Amino Acid Supplementation in Older Adult COVID-19 Patients
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: PI no longer wanted to do the study
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 261678
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2021-05

CONDITIONS: Covid19
Keywords: Amino acid supplement; Dietary supplement
MeSH Terms: conditions — COVID-19 | interventions — Amino Acids, Essential; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- EAA - non-vaccinated (Experimental): 18 g/day
  Interventions: Drug: Essential amino acids
- Placebo - non-vaccinated (Placebo Comparator): 18 g/day
  Interventions: Dietary Supplement: Maltodextrin
- EAA - vaccinated (Experimental): 18 g/day
  Interventions: Drug: Essential amino acids
- Placebo - vaccinated (Placebo Comparator): 18 g/day
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Drug: Essential amino acids — Dietary Supplement
  Other Names: EAA
  Arms: EAA - non-vaccinated; EAA - vaccinated
Dietary Supplement: Maltodextrin — Control
  Arms: Placebo - non-vaccinated; Placebo - vaccinated

SUMMARY:
A 4-week treatment of essential amino acids or placebo to participants with: 1) negative COVID-19 test with exposure, or 2) positive COVID-19 test and no or mild symptoms. The study team will measure change in symptoms. Participants will complete symptom surveys for 4 weeks and once at 8 and 12 weeks as well as pre- and post-assessments.

DETAILED DESCRIPTION:
In people who have been exposed to COVID-19 and have been tested (positive or negative) with no to mild symptoms, the study team will administer a treatment of essential amino acids (EAA). The study team will examine if this treatment compared to placebo will reduce the development, length and the severity of symptoms. Participants will consume the treatment or placebo for 4 weeks, and will complete symptom surveys, as well as pre- and post-assessments. Individuals who receive a COVID vaccination will continue to complete symptom surveys for 1 week and take the essential amino acid supplementation for 2 weeks following a vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Exposure to COVID-19 in the last 60 days with no symptoms, with a COVID negative test Close contact: within 6 feet of a COVID-19 positive person for more than a few minutes without wearing PPE, or having direct contact with infectious secretions without PPE
* Positive COVID-19 test with or without symptoms

Exclusion Criteria:

* COVID-19 positive hospitalized patient
* Patients who have symptoms of COVID but have not been tested.
* Unable to tolerate oral intake
* In hospice or palliative care
* Unstable medical or psychiatric condition
* Other criteria deemed acceptable by principle investigator

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Improvement in symptoms | 12 weeks
  Decrease in EAA group symptom score compared to placebo by 25%

CONTACTS AND LOCATIONS:
Overall Officials: Gohar Azhar, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No